CLINICAL TRIAL: NCT02801617
Title: A Multicentric, Prospective, Crossover, Double Blind Clinical Study to Evaluate the Non-inferiority of PRO-067 an Ophthlamic Solution Manufactured by Laboratorios Sophia S.A.de C.V., Previous Treatment With GAAP Ofteno ®, in Subjects With Primary Open-angle Glaucoma (POAG) or Ocular Hypertension (OHT): COMPLIANCE Study
Brief Title: Non-inferiority of PRO-067 Ophthalmic Solution vs GAAP Ofteno® in Glaucoma or Ocular Hypertension
Acronym: COMPLIANCE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: expiration time limit of recruitment
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH067-0914/III
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Latanoprost; Glaucoma; Ocular hypertension; Crossover study
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Latanoprost; Prostaglandins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (PRO-067) (Experimental): study subjects will be allocated to receive PRO-067 QD for 30 days, after which they will be crossed over to the other medication (GAAP Ofteno®) for another 30 days. The Intraocular pressure-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline.
  Washout period: 21 hours
  Interventions: Drug: PRO-067; Drug: GAAP Ofteno®
- Sequence 2 (GAAP Ofteno®) (Active Comparator): study subjects will be allocated to receive GAAP Ofteno® QD for 30 days, after which they will be crossed over to the other medication (PRO-067) for another 30 days. The Intraocular pressure-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline.
  Washout period: 21 hours
  Interventions: Drug: PRO-067; Drug: GAAP Ofteno®

INTERVENTIONS:
Drug: PRO-067 — 1 drop QD during 30 days is a sterile ophthalmic solution formulated by Laboratorios Sophia S.A. de C.V.
  Other Names: SOPH067-0914/III
Drug: GAAP Ofteno® — 1 drop QD during 30 days Active comparator, reference medication.
  Other Names: Latanoprost 0.005% , prostaglandin, antiglaucoma medication

SUMMARY:
Aim: To demonstrate the non-inferiority of the PRO-067 ophthalmic solution manufactured by Laboratorios Sophia S.A. de C.V. versus GAAP Ofteno® ophthalmic solution like hypotensive therapy in subjects with primary open angle glaucoma or ocular hypertension.

Study design: a multicentric, prospective, crossover (2x2), double blind clinical study. Sample size: one hundred patients with primary open angle glaucoma or ocular hypertension. Patients in the period 1: In the first sequence 60 patients will be assigned to receive the ophthalmic solution: GAAP Ofteno ® (latanoprost 0.005%) 1 drop per day (QD) during 30 days and the second sequence 60 patients will be assigned to receive the ophthalmic solution: PRO-067 1 drop QD during 30 days in the same period. Washout period: 21 hours. Patients in the period 2: the pharmacological intervention change to the opposite therapy for 30 days.

DETAILED DESCRIPTION:
The American Academy of Ophthalmology Glaucoma Panel The primary open angle glaucoma (POAG) is a progressive, chronic optic neuropathy in adults in which intraocular pressure (IOP) and other currently unknown factors contribute to damage and in which, in the absence of other identifiable causes, there is a characteristic acquired atrophy of the optic nerve and loss of retinal ganglion cells and their axons. This condition is associated with an anterior chamber angle that is open by gonioscopic appearance.

This is a multicentric, crossover, double blind and prospective clinical study. The investigators will include patients with confirmed diagnosis of primary open-angle glaucoma or ocular hypertension, with target intraocular pressure (TIOP) within a range at which a patient is likely to remain stable or at which worsening of glaucoma will be slow enough that the risk of additional intervention is not justified.

Patients will be randomly divided into 2 groups, one of them treated with a known formulation of Latanoprost 0.005% (GAAP Ofteno®, Laboratorios Sophia, Mexico) and the other one treated with PRO-067 ophthalmic solution. Patients will receive 1 drop per day (QD) into the lower conjunctival sac of either formulations and were examined at days: 1, 15, 30, 45 ad 60 after initiation of treatment. A phone call security at day 75 will be performed.

Primary efficacy outcome: To evaluate the efficacy of PRO-067 versus GAAP Ofteno ® instilled onto the ocular surface in subjects with primary open angle glaucoma (POAG) or ocular hypertension (HTO), to control and maintenance of the target intraocular pressure (TIOP).

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* Age: ≥18 years old
* Patients with primary open angle glaucoma with mild to moderate damage or ocular hypertension that were sufficiently controlled with GAAP Ofteno® (latanoprost 0.005%) within the last 60 days
* Signed Informed Consent Form

Exclusion Criteria:

* Subjects with unique eye
* Subjects with visual acuity < 20/200
* Another kind of glaucoma disease different to primary open angle glaucoma
* corneal disturbances with impossibility to measure the intraocular pressure
* retinal alterations without control or progressive retinal disease with high risk to lost vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03-15 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Contract Research Organization, Zapopan, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
Electronic Case Report Format (eCRF). The on line registry in a digital platform will help to verification process.

REFERENCES:
- See also: Mexican Registry of Clinical trials. The Federal Commission for the Protection against Sanitary Risk (COFEPRIS) — http://189.254.115.250/Resoluciones/Consultas/ConWebRegEnsayosClinicosDetalle.asp?idsolicitud=2036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study raised 120 research subjects, only 116 were selected, 2 left the study before being evaluated for a total of 114. However, 7 subjects were eliminated by: closure of center 1, without monitoring 2, by loss of follow-up 2, non-compliance with inclusion criteria 1 and failure of scrutiny 1, leaving a total of 107 randomized research subjects
Groups:
- Sequence 1 (PRO-067): study subjects will be allocated to receive PRO-067 QD for 30 days, after which they will be crossed over to the other medication (GAAP Ofteno®) for another 30 days. The Intraocular pressure-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline.
  Washout period: 21 hours
  PRO-067: 1 drop QD during 30 days is a sterile ophthalmic solution formulated by Laboratorios Sophia S.A. de C.V.
  GAAP Ofteno®: 1 drop QD during 30 days Active comparator, reference medication.
- Sequence 2 (GAAP Ofteno®): study subjects will be allocated to receive GAAP Ofteno® QD for 30 days, after which they will be crossed over to the other medication (PRO-067) for another 30 days. The Intraocular pressure-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline.
  Washout period: 21 hours
  PRO-067: 1 drop QD during 30 days is a sterile ophthalmic solution formulated by Laboratorios Sophia S.A. de C.V.
  GAAP Ofteno®: 1 drop QD during 30 days Active comparator, reference medication.
Period: Overall Study
Arm/Group | Sequence 1 (PRO-067) | Sequence 2 (GAAP Ofteno®)
Started | 51 | 56
Completed | 49 | 50
Not Completed | 2 | 6
Not completed — Protocol Violation | 2 | 6

BASELINE CHARACTERISTICS:
Population: the estadistic analysis was performed by protocol for the primary variable and by intention to treat in tolerability and adverse events.
Groups:
- Sequence 1 (PRO-067): 60 study subjects will be allocated to receive PRO-067 QD for 30 days, after which they will be crossed over to the other medication (GAAP Ofteno®) for another 30 days. The Intraocular pressure-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline.
  Washout period: 21 hours
  PRO-067: 1 drop QD during 30 days is a sterile ophthalmic solution formulated by Laboratorios Sophia S.A. de C.V.
  GAAP Ofteno®: 1 drop QD during 30 days Active comparator, reference medication.
- Sequence 2 (GAAP Ofteno®): 60 study subjects will be allocated to receive GAAP Ofteno® QD for 30 days, after which they will be crossed over to the other medication (PRO-067) for another 30 days. The Intraocular pressure-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline.
  Washout period: 21 hours
  PRO-067: 1 drop QD during 30 days is a sterile ophthalmic solution formulated by Laboratorios Sophia S.A. de C.V.
  GAAP Ofteno®: 1 drop QD during 30 days Active comparator, reference medication.
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (PRO-067) | Sequence 2 (GAAP Ofteno®) | Total
Number analyzed (Participants) | 51 | 56 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 62
  >=65 years | 21 | 24 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 47 | 83
  Male | 15 | 9 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 51 | 56 | 107

OUTCOME MEASURES:

1. Primary Outcome: Target Intraocular Pressure (TIOP)
Description: Target Intraocular Pressure (TIOP): Efficacy of experimental drug or active comparator to maintain the IOP in a range at which a patient is likely to remain stable or at which worsening of glaucoma will be slow enough that the risk of additional intervention is not justified.The upper limit of intraocular pressure is: TIOP + 2 mmHg. The measurement of the TIOP in each treatment period.
Time Frame: the baseline visit (day 0), Cross Over Visit (day 30) and the final visit (day 60) for both sequences
Population: by Protocol
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Sequence A (PRO-067- GAAP Ofteno®): First Period. PRO-067: 1 drop QD (per day) during 30 days is a sterile ophthalmic solution formulated by Laboratorios Sophia S.A. de C.V.
  Second period. GAAP Ofteno®: 1 drop QD during 30 days Active comparator, reference medication.
- Sequence B (GAAP Ofteno® - PRO-067): Fist Period. GAAP Ofteno®: 1 drop QD (per day) during 30 days Active comparator, reference medication.
  Second Period. PRO-067: 1 drop QD during 30 days is a sterile ophthalmic solution formulated by Laboratorios Sophia S.A. de C.V.
Arm/Group | Sequence A (PRO-067- GAAP Ofteno®) | Sequence B (GAAP Ofteno® - PRO-067)
Number analyzed (Participants) | 49 | 50
mmHg
  baseline visit | 14.25 (2.37) | 14.04 (2.43)
  Cross over visit | 13.85 (2.07) | 13.92 (2.17)
  final visit | 13.99 (2.46) | 14.07 (2.37)
Statistical Analysis 1: Comparison: Sequence A (PRO-067- GAAP Ofteno®); Test type: Non-Inferiority — it will be considered not inferior if they keep the IOP goal with differences of no more than 2 mmHg analysis by protocol; p = 0.861, t-test, 2 sided
Statistical Analysis 2: Comparison: Sequence B (GAAP Ofteno® - PRO-067); Test type: Non-Inferiority — it will be considered not inferior if they keep the TIOP with differences of no more than 2 mmHg; p = 0.890, t-test, 2 sided

2. Primary Outcome: Number of Adverse Events.
Description: the two periods of PRO-067 of each sequence were grouped as well as those of GAAP to form two comparative groups of adverse events in each intervention. (PRO-067 vs. GAAP ofteno).
  The number of adverse events presented throughout the study was evaluated with each study drug to make the comparison between groups.
Time Frame: it is evaluated from the baseline visit (day 1) to the security call (day 75)
Population: intention-to-treat (ITT), all those subjects who received at least one dose of the investigational drugs were considered for the statistical analysis, having a total of 107 cases by intention to treat.
Measure: Number; unit: adverse events
Groups:
- PRO-067: PRO-067,QD (per day) for 60 days. Includes both periods of PRO-067 in sequence A and B.
- GAAP Ofteno®: GAAP Ofteno® QD (per day) for 60 days. Includes both periods of GAAP in sequence A and B.
Arm/Group | PRO-067 | GAAP Ofteno®
Number analyzed (Participants) | 51 | 56
adverse events | 24 | 20
Statistical Analysis 1: Comparison: PRO-067 vs GAAP Ofteno®; Test type: Non-Inferiority — intention-to-treat analysis (ITT); p = 0.329, Chi-squared

3. Secondary Outcome: Percentage of Ocular Burning
Description: the ocular burning of the study subjects was evaluated, during the baseline, crossover and final visit, the variable was described as present or absent, according to the case, in both groups. A Pearson´s chi-square test is performed in the crossover and final visit to compare the end of periods 1 and 2 between both study sequences.
Time Frame: at the basal visit (day 1) crossover visit (day 30) and final visit (day 60)
Population: analysis by protocol
Measure: Number; unit: percentage of Ocular burning
Groups:
- Sequence 1 (PRO-067): Study subjects will be allocated to receive:
  PRO-067: 1 drop QD (per day) during 30 days after GAAP Ofteno®: 1 drop QD during 30 days
- Sequence 2 (GAAP Ofteno®): Study subjects will be allocated to receive:
  GAAP Ofteno®: 1 drop QD (per day) during 30 days after PRO-067: 1 drop QD during 30 days
Arm/Group | Sequence 1 (PRO-067) | Sequence 2 (GAAP Ofteno®)
Number analyzed (Participants) | 49 | 50
percentage of Ocular burning
  basal visit | 20.7 | 19.6
  Crossover visit | 03.8 | 25.0
  Final visit | 10.3 | 16.1
Statistical Analysis 1: Comparison: Sequence 1 (PRO-067) vs Sequence 2 (GAAP Ofteno®); Test type: Non-Inferiority — it will be considered not inferior if they keep the percentage of ocular burning with differences of no more than 20%; p = 0.388, Chi-squared, Corrected

4. Secondary Outcome: Percentage of Participants With Foreign Body Sensation
Description: The foreign body sensation will be measured as present / absent according to each case. A Pearson´s chi-square test is performed in the crossover and final visit to compare the end of periods 1 and 2 between both study sequences.
Time Frame: basal visit (day 1), Crossover visit (day 30) and final visit (day 60)
Population: Analysis by protocol
Measure: Number; unit: percentage of patients with Foreign body
Arm/Group | Sequence A (PRO-067- GAAP Ofteno®) | Sequence B (GAAP Ofteno® - PRO-067)
Number analyzed (Participants) | 49 | 50
percentage of patients with Foreign body
  basal visit (day 1) | 20.7 | 37.5
  Crossover visit (day 30 | 24.1 | 30.4
  final visit (day 60) | 17.2 | 30.4
Statistical Analysis 1: Comparison: Sequence A (PRO-067- GAAP Ofteno®) vs Sequence B (GAAP Ofteno® - PRO-067); Test type: Non-Inferiority — it will be considered not inferior if they keep the percentage of ocular burning with differences of no more than 20%; p = 0.125, Chi-squared, Corrected

5. Secondary Outcome: Percentage of Participants With Tearing
Description: The tearing will be measured as present / absent according to each case. A Pearson´s chi-square test is performed in the crossover and final visit to compare the end of periods 1 and 2 between both study sequences.
Time Frame: basal visit (day 1), Crossover visit (day 30) and final visit (day 60)
Population: Analysis by protocol
Measure: Number; unit: percentage of patients with tearing
Arm/Group | Sequence A (PRO-067- GAAP Ofteno®) | Sequence B (GAAP Ofteno® - PRO-067)
Number analyzed (Participants) | 49 | 50
percentage of patients with tearing
  Basal visit (day 1) | 8.6 | 5.4
  Crossover visit (day 30) | 8.6 | 10.7
  Final visit (day 60) | 3.4 | 7.1
Statistical Analysis 1: Comparison: Sequence A (PRO-067- GAAP Ofteno®) vs Sequence B (GAAP Ofteno® - PRO-067); Test type: Non-Inferiority — it will be considered not inferior if they keep the percentage of ocular burning with differences of no more than 20%; p = 0.434, Chi-squared, Corrected

6. Secondary Outcome: Percentage of Participants With Chemosis
Description: The chemosis will be measured as present / absent according to each case. A Pearson´s chi-square test is performed in the crossover and final visit to compare the end of periods 1 and 2 between both study sequences.
Time Frame: basal visit (day 1), Crossover visit (day 30) and final visit (day 60)
Population: Analysis by protocol
Measure: Number; unit: percentage of patients with chemosis
Arm/Group | Sequence A (PRO-067- GAAP Ofteno®) | Sequence B (GAAP Ofteno® - PRO-067)
Number analyzed (Participants) | 49 | 50
percentage of patients with chemosis
  basal visit (day 1) | 3.4 | 7.1
  Crossover visit (day 30) | 0 | 0
  final visit (day 60) | 0 | 0
Statistical Analysis 1: Comparison: Sequence A (PRO-067- GAAP Ofteno®) vs Sequence B (GAAP Ofteno® - PRO-067); Test type: Non-Inferiority — it will be considered not inferior if they keep the percentage of ocular burning with differences of no more than 20%; p = 0, Chi-squared, Corrected

7. Secondary Outcome: Percentage of Participants With Hyperemia
Description: the hyperemia of the study subjects was evaluated, during the baseline, crossover and final visit, the variable was described as a scale of: absent, very mild, mild, moderate and severe, according to the case, in both groups. A Pearson´s chi-square test is performed in the crossover and final visit to compare the end of periods 1 and 2 between both study sequences.
Time Frame: basal visit (day 1), Crossover visit (day 30) and final visit (day 60)
Population: Analysis by protocol
Measure: Number; unit: percentage of patients with hyperemia
Arm/Group | Sequence A (PRO-067- GAAP Ofteno®) | Sequence B (GAAP Ofteno® - PRO-067)
Number analyzed (Participants) | 49 | 50
percentage of patients with hyperemia
  Basal Visit Very Mild | 53.4 | 50.0
  Basal Visit Mild | 41.4 | 43.9
  Basal Visit Moderate | 5.2 | 4.4
  Cross Over Visit Very Mild | 60.3 | 51.8
  Cross Over Visit Mild | 37.9 | 44.6
  Cross Over Visit Moderate | 1.7 | 3.6
  Final visit Very Mild | 67.2 | 69.6
  Final Visit Mild | 32.8 | 23.2
  Final Visit Moderate | 0 | 7.1
Statistical Analysis 1: Comparison: Sequence A (PRO-067- GAAP Ofteno®) vs Sequence B (GAAP Ofteno® - PRO-067); Test type: Non-Inferiority — it will be considered not inferior if they keep the percentage of ocular burning with differences of no more than 20%; p = 0.039, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during 75 days, from the baseline visit (day 1) to the safety call (day 75)
Groups:
- PRO-067: PRO-067,QD for 60 days. Includes both periods of PRO-067 in sequence A and B.
- GAAP Ofteno®: GAAP Ofteno®, QD for 60 days. Includes both periods of PRO-067 in sequence A and B.
Arm/Group | PRO-067 | GAAP Ofteno®
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/56
Other Adverse Events (participants affected / at risk) | 24/51 | 20/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-067 (N=51) | GAAP Ofteno® (N=56)
Conjuntivitis (Eye disorders) | 2 (2) | 5 (5)
itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 3 (3) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
rhinopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
headache (General disorders) | 3 (3) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
subconjunctival hemorrhage (Eye disorders) | 1 (1) | 3 (3)
Sleep disorder (General disorders) | 1 (1) | 0 (0)
arterial hypertension (Vascular disorders) | 1 (1) | 1 (1)
ankle bruise (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dental process (Gastrointestinal disorders) | 0 (0) | 2 (2)
spasm orbicularis oculi (Eye disorders) | 1 (1) | 0 (0)
hypercholesterolemia (Endocrine disorders) | 0 (0) | 1 (1)
venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations of this study were its short duration (60 days) and the size of the groups that was reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT02801617/Prot_SAP_000.pdf